CLINICAL TRIAL: NCT04523220
Title: A Randomized, Double-blind, Parallel Group, Placebo-controlled, Multi-center Study to Assess the Safety and Tolerability of Monthly Subcutaneous Administrations of a Low and High Dose Cohort of Osocimab to ESRD Patients on Regular Hemodialysis
Brief Title: Study to Investigate the Safety of a Drug Called Osocimab at Low and High Doses in Adult Patients With Kidney Failure Requiring Regular Hemodialysis
Acronym: CONVERT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20115; 2019-003957-27 (EudraCT Number)
Record Dates: First submitted 2020-08-20; First posted 2020-08-21 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: End-stage Renal Disease; Prevention of Thromboembolic Events; Hemodialysis; Hemodiafiltration
Keywords: End-stage renal disease (ESRD); Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — osocimab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BAY1213790 low dose (Experimental): Participants will receive Osocimab (BAY1213790) 105 mg single loading dose as subcutaneous abdominal injection, followed by monthly maintenance doses of 52.5 mg until the end of the extension treatment period.
  Interventions: Drug: BAY1213790 (Osocimab)
- Placebo low dose (Placebo Comparator): Placebo will be administered subcutaneously in the same manner as Osocimab.
  Interventions: Drug: Placebo
- BAY1213790 high dose (Experimental): Participants will receive Osocimab (BAY1213790) 210 mg single loading dose as subcutaneous abdominal injection, followed by monthly maintenance doses of 105 mg until the end of the extension treatment period.
  Interventions: Drug: BAY1213790 (Osocimab)
- Placebo high dose (Experimental): Placebo will be administered subcutaneously in the same manner as Osocimab.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY1213790 (Osocimab) — Single loading dose as subcutaneous abdominal injection followed by monthly maintenance doses.
  Arms: BAY1213790 high dose; BAY1213790 low dose
Drug: Placebo — Subcutaneous administration in the same manner as Osocimab.
  Arms: Placebo high dose; Placebo low dose

SUMMARY:
In this study researchers want to learn about the safety of drug Osocimab at lower-dose and higher-doses in adult participants with kidney disease undergoing regular dialysis (a procedure that uses a machine to get rid of toxins and extra fluids in the blood). Patients with kidney disease undergoing regular dialysis are at high risk for heart and blood vessels diseases. Osocimab is a human monoclonal antibody under development for the prevention of events caused by blood clots like heart attack, stroke and death due to heart or blood vessels diseases. It works by binding to and blocking the activated form of clotting factor XI which increases the formation and stability of clots. Researchers also want to find out how drug Osocimab works in human body and how the body absorbs, distributes and excretes the drug.

Participants in this study will receive monthly injection of either Osocimab at a lower-dose or higher-dose or placebo (a placebo looks like a treatment but does not have any medicine in it). Both Osocimab and placebo will be injected into the tissue under the skin of the belly. Observation for each participant will last up to 23 months. Blood samples will be collected from the participants to monitor the safety and measure the blood level of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age
* Patients with end-stage renal disease on hemodialysis (including hemodiafiltration) for ≥3 months, receiving dialysis at least 9 hours a week and stable in the view of the investigator
* Body weight of at least 50 kg
* Male and/or female. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Recent (<6 months before screening) clinically significant bleeding
* Hemoglobin (Hb) < 9.0 g/dL at screening
* Platelet count < 100 x 10^9/L
* aPTT or PT > ULN (upper limit of normal)
* Hepatic disease associated with ALT > 3x ULN, or total bilirubin >2x ULN with direct bilirubin > 20% of the total
* Sustained uncontrolled hypertension (diastolic blood pressure ≥100 mmHg and/or systolic blood pressure ≥ 180 mmHg)
* Known intracranial neoplasm, arteriovenous malformation or aneurysm
* Known bleeding disorders e.g. von-Willebrand disease or Hemophilia A, B or C
* Recent (<3 months before screening) thromboembolic event, e.g. acute coronary syndrome, stroke or VTE (except dialysis access thrombosis)
* Recent (<3 months before screening) major surgery or scheduled major surgery during study participation
* Scheduled living donor renal transplant during study participation
* Persistent heart failure as classified by the New York Heart Association (NYHA) classification of 3 or higher
* Receiving antiplatelet therapy except daily ASA ≤ 150 mg/day
* Receiving anticoagulation in therapeutic doses, other than standard anticoagulation during the hemodialysis procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 704 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2022-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (151):
- United States (26):
  - North America Research Institute - Azusa, Azusa, California
  - Fresenius Kidney Care - Brawley, Brawley, California
  - DaVita South Valley Dialysis, Encino, California
  - Fresenius Kidney Care - La Mesa, La Mesa, California
  - East L.A. Dialysis Center, Los Angeles, California
  - Van Buren Dialysis Center, Riverside, California
  - Fresenius Kidney Care Kearny Mesa, San Diego, California
  - FMC San Ysidro, San Diego, California
  - Queen's Dialysis Unit, West Covina, California
  - DaVita Greater Waterbury Dialysis, Waterbury, Connecticut
  - ARA Plantation Dialysis, LLC, Ellenton, Florida
  - ARA Augusta, Augusta, Georgia
  - Liberty Dialysis- Caldwell, Caldwell, Idaho
  - Fresenius Kidney Care Evergreen Park, Evergreen Park, Illinois
  - Fresenius Kidney Care Baton Rouge Mancuso Lane, Baton Rouge, Louisiana
  - Fresenius Kidney Care South Dialysis, Shreveport, Louisiana
  - ARA Holyoke Dialysis Center, Holyoke, Massachusetts
  - Davita Hospital Hill Dialysis, Kansas City, Missouri
  - Renal Medicine Associates, Albuquerque, New Mexico
  - Durham Nephrology Associates, Pa, Durham, North Carolina
  - Waterloo Dialysis, Austin, Texas
  - Fresenius North Austin Dialysis Center, Austin, Texas
  - Fresenius Kidney Care - Mission Bend (FMCNA #3971), Houston, Texas
  - Fresenius Kidney Care Sugar Land, Sugar Land, Texas
  - Liberty Dialysis St. George, St. George, Utah
  - DaVita Butler Farm Dialysis, Hampton, Virginia
- Australia (4):
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Eastern Health Integrated Renal Service, Box Hill
  - John Hunter Hospital, New Lambton Heights
- Austria (4):
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt, Carinthia
  - Privatklinik Wehrle-Diakonissen, Salzburg
  - Klinik Landstraße - Krankenhaus Rudolfstiftung, Vienna
  - Universitätsklinikum AKH Wien, Vienna
- Belgium (6):
  - Epicura, Baudour
  - Imeldaziekenhuis - St-Elisabethkliniek, Bonheiden
  - AZ St-Lucas Campus St-Lucas, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - CHU de Liege | CHR Citadel - Department of Nephrology, Liège
  - AZ Nikolaas Campus Sint-Niklaas, Sint-Niklaas
- Bulgaria (5):
  - MHAT Sveti Ivan Rilski 2003, Dupnitsa
  - MHAT Haskovo, Haskovo
  - UMHAT Kanev AD, Rousse
  - MHAT Shumen AD, Shumen
  - Multiprofile Hospital for Active Treatment Hristo Botev AD, Vratsa
- Czechia (4):
  - Krajska Nemocnice Liberec, Liberec
  - Fakultni nemocnice Ostrava, Ostrava
  - Privamed s.r.o., Pilsen
  - Fresenius Nephro Care s.r.o. - Sokolov, Sokolov
- Greece (7):
  - General Hospital of Arta, Arta
  - HIPPOKRATION General Hospital of Athens, Athens
  - General Hospital of Athens LAIKO, Athens
  - Ioannina University General Hospital, Ioannina
  - University General Hospital of Larissa, Larissa
  - Hippokration General Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki Papageorgiou, Thessaloniki
- Hungary (7):
  - Bajai Szent Rokus Korhaz, Baja
  - Fresenius Medical Care Egeszsegugyi Kft., Budapest
  - Eszak-Pesti Centrumkorhaz-Honvedkorhaz, Budapest
  - Csongrad Megyei Egeszsegugyi Ellato Kozpont,Hodmezovasarhely, Hódmezővásárhely
  - Keszthelyi Korhaz, Keszthely
  - Fresenius Medical Care Egeszsegugyi Kft., Miskolc
  - Fresenius Medical Care Egeszsegugyi Kft., Pécs
- Israel (7):
  - Barzilai Medical Center | Nephrology & Hypertension Dept., Ashkelon
  - Lady Davis Carmel Medical Center, Haifa
  - Health Corporation of Galilee Medical Center, Nahariya
  - Rabin Medical Center, HaSharon (Golda) Campus, Petah Tikva
  - Clalit Health Services Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Poriya Medical Center | Nephrology and Hypertension Dept., Tiberius
  - Shamir Medical Center (Assaf Harofeh), Ẕerifin
- Italy (7):
  - A.O.U. di Bologna Policlinico S.Orsola Malpighi, Bologna, Emilia-Romagna
  - A.O.U. di Parma, Parma, Emilia-Romagna
  - AUSL-IRCCS di Reggio Emilia, Reggio Emilia, Emilia-Romagna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - IRCCS Ospedale Policlinico San Martino, Genoa, Liguria
  - IRCCS Istituti Clinici Scientifici Maugeri SpA SB, Pavia, Lombardy
  - A.O.U. Careggi, Florence, Tuscany
- Japan (14):
  - Ibaraki Seinan Medical Center Hospital, Sashima-gun, Ibaraki
  - Tsuchiura Beryl Clinic, Tsuchiura, Ibaraki
  - Ohishi Naika Clinic, Tsuchiura, Ibaraki
  - Kikuchi Medical Clinic, Tsukuba, Ibaraki
  - Katta General Hospital, Shiraishi, Miyagi
  - Nagaoka Red Cross Hospital, Nagaoka, Niigata
  - Saiyu Clinic, Koshigaya, Saitama
  - Takemura Medical Nephro Clinic, Kanuma, Tochigi
  - Futakotamagawaekimae clinic, Setagaya-ku, Tokyo
  - Saint Hill Hospital, Ube, Yamaguchi
  - Akebono Clinic, Kumamoto
  - Kyoto Station Takeda Dialysis Clinic, Kyoto
  - Akagaki Clinic, Osaka
  - Yabuki Hospital, Yamagata
- LUHS Kauno Hospital (Josvainiu str.), Kaunas, Lithuania
- Netherlands (6):
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Deventer Ziekenhuis, Deventer
  - Albert Schweitzer Ziekenhuis, Dordwijk, Dordrecht
  - Catharina Ziekenhuis, Eindhoven
  - Maasstad Ziekenhuis | Neurology Department, Rotterdam
- Poland (5):
  - NZOZ Nowy Szpital w Swieciu Sp. z o.o., Gmina Świecie
  - Wojewodzki Szpital Zespolony, Kielce
  - Stacja Dializ Olkusz, Olkusz
  - Stacja Dializ W-wa Mangalia, Warsaw
  - Stacja Dializ Zyrardow, Żyrardów
- Portugal (10):
  - Eurodial Obidos (DaVita), Gaeiras - Obidos, Leiria District
  - SPD - Amadora (Diaverum Amadora), Amadora, Lisbon District
  - CHLO - Hospital Santa Cruz, Carnaxide, Lisbon District
  - Pluribus Dialise - Cascais (DaVita), Cascais, Lisbon District
  - Pluribus Dialise - Sacavem (DaVita), Sacavém, Lisbon District
  - Caledial - Centro de Hemodialise de Gaia, Canelas, Porto District
  - Centro Hospitalar do Medio Tejo | Unidade de Torres Novas - Nephrology Department, Torres Novas, Santarém District
  - Diaverum Aveiro, Aveiro
  - Eurodial Leiria (DaVita), Leiria
  - NephroCare APDP, Lisbon
- Russia (11):
  - Chelyabinsk Regional Clinical Hospital, Chelyabinsk
  - LLC Dialysis center, Kolomna
  - LLC Fresenius medical care Kuban, Krasnodar
  - LLC Dialysis center, Mytishchi
  - City Clinical Hospital #1 Orenburg, Orenburg
  - Republican Hospital n.a. V.A. Baranov, Petrozavodsk
  - Kupchinsky center for outpatient dialysis, Saint Petersburg
  - LLC B. Brown Avitum Russland Clinics, Saint Petersburg
  - City Hospital #31, Saint Petersburg
  - LLC Yaroslavl dialysis center, Yaroslavl
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- Spain (7):
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Althaia, Xarxa Assistencial de Manresa, Manresa, Barcelona
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital Clinico Universitario San Carlos | Nefrologia, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
- Turkey (Türkiye) (7):
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Adnan Menderes Universitesi Tip fakultesi, Aydin
  - Turk Bobrek Vakfi Memorial Hizmet Hastanesi, Istanbul
  - Sisli Hamidiye Etfal Egitim ve Arastirma Hastanesi, Istanbul
  - Erciyes Universitesi Tip Fakultesi, Kayseri
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Inonu Universitesi Tip Fakultesi, Malatya
- Ukraine (13):
  - Brovarskaya multidisciplinary clinical hospital, Brovary
  - Medical center LLC " Fresenius medical care Ukraine", Cherkasy
  - Dnepropetrovsk regional hospital n.a. I. I. Mechnikov, Dnipro
  - Regional Clinical Hospital - Ivano-Frankivsk, Ivano-Frankivsk
  - Kharkiv regional Clinical Centre of urology and nephrology, Kharkiv
  - Kyiv City Center of Nephrology and Dialysis, Kyiv
  - State Institution "Institute of Nephrology" NAMS of Ukraine, Kyiv
  - Lutsk city clinical hospital, Lutsk
  - Mykolaiv Regional Clinical Hospital, Mykolaiv
  - Poltava Regional Clinical Hospital n.a. M.V. Skliphosovskyi, Poltava
  - Transcarpatian Regional Clinical Hospital, Uzhhorod
  - Vinnitsa Regional Clinical Hospital im. N.I. Pirogov, Vinnytsia
  - Zaporizhzhia Regional Clinical Hospital, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share data.

REFERENCES:
- [Derived] Weitz JI, Tanko LB, Floege J, Fox KAA, Bhatt DL, Thadhani R, Hung J, Pap AF, Kubitza D, Winkelmayer WC; CONVERT Investigators. Anticoagulation with osocimab in patients with kidney failure undergoing hemodialysis: a randomized phase 2 trial. Nat Med. 2024 Feb;30(2):435-442. doi: 10.1038/s41591-023-02794-7. Epub 2024 Feb 16. PMID 38365952
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in 19 countries/regions, between 28-Aug-2020 (first participant first visit) and 30-May-2022 (last participant last visit).
Pre-assignment Details: A total of 859 participants were screened; 155 participants were not randomized. Most common reason for not being randomized was screen failure (144 participants). 704 participants were randomized to treatment; 18 participants did not receive treatment. The remaining 686 participants were treated.
Groups:
- Higher-dose Osocimab: Participants were randomized to receive Osocimab (BAY1213790) 210 mg single loading dose as subcutaneous abdominal injection, followed by monthly maintenance doses of 105 mg for 6 months in main treatment phase.
  Participants received Osocimab (BAY1213790) at monthly maintenance doses of 105 mg up to a maximum of 12 months or until the last participant randomized to the study has performed the end of main treatment (EOMT) visit (whichever comes first) in extension treatment period.
- Lower-dose Osocimab: Participants were randomized to receive Osocimab (BAY1213790) 105 mg single loading dose as subcutaneous abdominal injection, followed by monthly maintenance doses of 52.5 mg for 6 months in main treatment phase.
  Participants received Osocimab (BAY1213790) at monthly maintenance doses of 52.5 mg up to a maximum of 12 months or until the last participant randomized to the study has performed the end of main treatment (EOMT) visit (whichever comes first) in extension treatment period.
- Placebo: Participants were randomized to receive matching placebo subcutaneously in the same manner as Osocimab.
Period: Main Treatment Period
Arm/Group | Higher-dose Osocimab | Lower-dose Osocimab | Placebo
Started (Randomized) | 234 | 235 | 235
Treated | 224 | 232 | 230
Completed | 194 | 199 | 206
Not Completed | 40 | 36 | 29
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Other | 5 | 2 | 4
Not completed — Subject Decision | 5 | 7 | 3
Not completed — Death | 5 | 11 | 4
Not completed — Adverse Event | 11 | 9 | 9
Not completed — Withdrawal by Subject | 3 | 3 | 4
Not completed — Study drug never adminstered | 10 | 3 | 5
Period: Extension Treatment Period
Arm/Group | Higher-dose Osocimab | Lower-dose Osocimab | Placebo
Started | 194 | 199 | 206
Completed | 174 | 178 | 176
Not Completed | 20 | 21 | 30
Not completed — Physician Decision | 1 | 0 | 3
Not completed — Other | 2 | 6 | 6
Not completed — Subject Decision | 5 | 2 | 4
Not completed — Death | 6 | 4 | 7
Not completed — Adverse Event | 6 | 7 | 9
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Study drug never administered | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: FAS (full analysis set): All participants randomly assigned to study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Higher-dose Osocimab | Lower-dose Osocimab | Placebo | Total
Number analyzed (Participants) | 234 | 235 | 235 | 704
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (13.4) | 61.1 (12.9) | 59.5 (13.3) | 60.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 90 | 81 | 256
  Male | 149 | 145 | 154 | 448
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 21 | 21 | 21 | 63
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 19 | 18 | 22 | 59
  White | 193 | 194 | 190 | 577
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Activated partial thromboplastin time (aPTT) value at baseline [Geometric Mean (Standard Deviation); unit: seconds] — aPTT was measured via the kaolin-trigger method (clotting assay). Furthermore, the aPTT assay was conducted after in vitro- neutralization of heparin in order to separate potential heparin effects from the PD effect of osocimab. Population: Participants in PDS with evaluable assessment for this measurement.
  seconds
    number analyzed (Participants) | 209 | 213 | 206 | 628
    (all) | 31.49 (1.10) | 31.32 (1.10) | 31.65 (1.09) | 31.49 (1.09)
Factor XI (FXI) activity at baseline [Geometric Mean (Standard Deviation); unit: percent] — Factor XI activity was assessed with an aPTT-based coagulation test using FXI deficient plasma. Furthermore, the assay was conducted after in vitro-neutralization of heparin in order to separate potential heparin effects from the PD effect of osocimab. Population: Participants in PDS with evaluable assessment for this measurement.
  percent
    number analyzed (Participants) | 208 | 212 | 202 | 622
    (all) | 100.54 (1.29) | 102.27 (1.28) | 103.09 (1.25) | 101.96 (1.27)

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence Risk of the First Composite of Major Bleeding (MB) and Clinically-relevant Non-major Bleeding (CRNMB) Events as Assessed by Blinded Central Independent Adjudication Committee (CIAC)
Description: Cumulative incidence risk of the first Composite of MB and CRNMB (ISTH) at month 6 is reported in the table.
  Descriptive time to composite of MB and CRNMB Events is reported in statistical analysis.
  Descriptive time to composite of treatment emergent major and CRNMB events [in alignment with International Society on Thrombosis and Haemostatsis (ISTH) guidelines] analyses were performed. The cumulative incidence function for the event-of-interest together with the corresponding confidence interval were estimated for each treatment arm using Aalen-Johansen estimators. Cumulative incidence of events up to the day, inclusive.
Time Frame: From the first dose of study intervention up till 30 days after last study intervention in the main treatment period, up to 6 months
Population: SAF (Safety analysis set): All participants randomly assigned to study intervention who took at least 1 dose of study intervention. Participants were analyzed according to the intervention they actually received.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Higher-dose Osocimab | Lower-dose Osocimab | Placebo
Number analyzed (Participants) | 224 | 232 | 230
Percentage of participants | 3.57 [1.91 to 6.04] | 4.32 [2.48 to 6.91] | 6.09 [3.84 to 9.04]
Statistical Analysis 1: Comparison: Higher-dose Osocimab vs Placebo; Two-sided log-rank tests and Cox proportional hazards model were used in the analyses; Test type: Other; p = 0.222, Log Rank — Due to the explorative nature of these analyses, no multiplicity adjustment was done; Cox Proportional Hazard = 0.59, 90% CI 2-sided [0.28 to 1.21]
Statistical Analysis 2: Comparison: Lower-dose Osocimab vs Placebo; Two-sided log-rank tests and Cox proportional hazards model were used in the analyses; Test type: Other; p = 0.427, Log Rank — Due to the explorative nature of these analyses, no multiplicity adjustment was done; Cox Proportional Hazard = 0.72, 90% CI 2-sided [0.36 to 1.42]

2. Primary Outcome: Cumulative Incidence Risk of Composite of Moderate and Severe Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Cumulative incidence risk of composite of moderate and severe AEs and SAEs at month 6 is reported in the table.
  Descriptive time to the composite of Moderate and Severe AEs and SAEs is reported in statistical analysis.
  An AE was any untoward medical occurrence in a patient or clinical study participant, whether or not considered related to the study intervention.
Time Frame: From the first dose of study intervention up until 30 days after last study intervention in the main treatment period, up to 6 months
Population: SAF (Safety analysis set)
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Higher-dose Osocimab | Lower-dose Osocimab | Placebo
Number analyzed (Participants) | 224 | 232 | 230
Percentage of participants | 38.84 [33.46 to 44.17] | 38.37 [33.10 to 43.60] | 32.17 [27.16 to 37.28]
Statistical Analysis 1: Comparison: Higher-dose Osocimab vs Placebo; Two-sided log-rank tests and Cox proportional hazards model were used in the analyses; Test type: Other; p = 0.128, Log Rank — Due to the explorative nature of these analyses, no multiplicity adjustment was done; Cox Proportional Hazard = 1.27, 90% CI 2-sided [0.98 to 1.64]
Statistical Analysis 2: Comparison: Lower-dose Osocimab vs Placebo; Two-sided log-rank tests and Cox proportional hazards model were used in the analyses; Test type: Other; p = 0.166, Log Rank — Due to the explorative nature of these analyses, no multiplicity adjustment was done; Cox Proportional Hazard = 1.24, 90% CI 2-sided [0.96 to 1.61]

3. Secondary Outcome: Ratio of Activated Partial Thromboplastin Time (aPTT) at 6 Months Trough Levels Versus Baseline.
Description: The aPTT at trough levels after 6 months were analyzed as ratio to baseline by providing the Geometric Mean (Standard Deviation).
  aPTT was measured via the kaolin-trigger method (clotting assay).
Time Frame: At 6 months (Visit 19 / Day 30 of the 6th month)
Population: PDS (Pharmacodynamic analysis set): All participants with at least 1 PD sample in accordance with the PD sampling schedule and without deviation from the protocol that would have interfered with the evaluation of the PD data were included in the PD analysis. Participants in PDS with data available for this outcome measure
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Higher-dose Osocimab | Lower-dose Osocimab | Placebo
Number analyzed (Participants) | 167 | 174 | 174
Ratio | 1.26 (1.11) | 1.19 (1.11) | 1.02 (1.08)

4. Secondary Outcome: Ratio of Factor XI (FXI) Activity at 6 Months Trough Levels Versus Baseline
Description: The Factor XI (FXI) activity at trough levels after 6 months were analyzed as ratio to baseline by providing the Geometric Mean (Standard Deviation).
  Factor XI activity was assessed with an aPTT-based coagulation test using FXI deficient plasma.
Time Frame: At 6 months (Visit 19 / Day 30 of the 6th month)
Population: PDS (Pharmacodynamic analysis set). Participants in PDS with data available for this outcome measure
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Higher-dose Osocimab | Lower-dose Osocimab | Placebo
Number analyzed (Participants) | 164 | 175 | 171
Ratio | 0.87 (1.27) | 0.94 (1.23) | 0.96 (1.20)

ADVERSE EVENTS:
Time Frame: After the first study intervention up until 30 days after last study intervention, with up to approximate 19 months. Adverse event reporting for the all-cause mortality considers all deaths that occurred at any time during the study before the last contact, with up to approximate 21 months.
Arm/Group | Higher-dose Osocimab | Lower-dose Osocimab | Placebo
All-Cause Mortality (participants affected / at risk) | 19/224 | 24/232 | 15/230
Serious Adverse Events (participants affected / at risk) | 61/224 | 67/232 | 63/230
Other Adverse Events (participants affected / at risk) | 90/224 | 85/232 | 88/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Higher-dose Osocimab (N=224) | Lower-dose Osocimab (N=232) | Placebo (N=230)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 2 (3) | 0 (0) | 1 (1)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperparathyroidism secondary (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal wall thickening (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0) | 4 (4)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Tuberculous pleurisy (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Febrile infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Renal cyst infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atypical mycobacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vascular access site infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 7 (7) | 8 (8) | 5 (5)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 9 (9) | 8 (8)
Device related bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Shunt occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Shunt stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Shunt aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1)
Unintentional medical device removal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access site inflammation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Angiocardiogram (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Nephrosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal haematoma (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal cyst ruptured (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Arteriovenous fistula operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Parathyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Renal transplant (Surgical and medical procedures) | 5 (5) | 3 (3) | 5 (5)
Toe amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Central venous catheterisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Dialysis device insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous graft (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Bladder neoplasm surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Peritoneal catheter insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 1 (2)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Iliac artery dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (2) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 1 (2)
Peripheral vein occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Higher-dose Osocimab (N=224) | Lower-dose Osocimab (N=232) | Placebo (N=230)
Anaemia (Blood and lymphatic system disorders) | 10 (10) | 12 (12) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 13 (16) | 6 (6) | 16 (18)
Vomiting (Gastrointestinal disorders) | 7 (7) | 8 (10) | 12 (16)
Pyrexia (General disorders) | 14 (15) | 9 (12) | 14 (17)
COVID-19 (Infections and infestations) | 11 (11) | 14 (14) | 12 (12)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 (20) | 9 (17) | 15 (23)
Headache (Nervous system disorders) | 19 (21) | 23 (26) | 14 (15)
Hypertension (Vascular disorders) | 18 (20) | 18 (24) | 16 (17)
Hypotension (Vascular disorders) | 15 (22) | 13 (27) | 18 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It's typically 30 days to review, and only if there is some need to file a patent application based on that review would there be an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT04523220/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT04523220/SAP_001.pdf